CLINICAL TRIAL: NCT02404636
Title: Alcohol Diet and Drug Use Preceding Alcoholic Hepatitis
Acronym: ADDUP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Birmingham (Other)
Responsible Party: Principal Investigator, Richard Parker, Clinical Lecturer, University Hospital Birmingham
Other Study IDs: RRK4357
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis, Alcoholic
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alcoholic hepatitis: Individuals admitted to hospital with acute alcoholic hepatitis, defined as acute onset of jaundice in the context of recent hazardous alcohol use and the absence of other liver disease
  Interventions: Other: Interview
- Hazardous alcohol use: Individuals admitted to hospital for any cause who drink hazardous quantities of alcohol but without evidence of alcoholic hepatitis or advanced liver disease
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Brief structured interview

SUMMARY:
ADDUP is an observational study of patients with alcoholic hepatitis. A structured interview is used to quantitatively estimate:

1. Alcohol use
2. Dietary intake
3. Drug use (legal and illegal)

in the weeks preceding onset of acute alcoholic hepatitis. After interview patients are followed up for 12 months with regard to response to therapy and survival.

The study is intended to explore potential precipitants of alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* acute alcoholic hepatitis
* aged over 18 years
* able to give informed consent

Exclusion Criteria:

* evidence of other acute or chronic liver disease
* episode of alcoholic hepatitis in 6 months before admission
* severe hepatic encephalopathy
* delirium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged over 18 years) admitted to Queen Elizabeth Hospital Birmingham, UK
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Changes in alcohol intake, dietary intake or drug use before illness | 1 month
  Behavior before admission (Brief structured interview)

SECONDARY OUTCOMES:
Survival after admission (Brief structured interview) | 12 months
  Survival
Response to treatment (Brief structured interview) | 1 week
  Response to treatment (corticosteroids, pentoxifylline or supportive medical care) after 1 week, measured by Lille score

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands, United Kingdom